CLINICAL TRIAL: NCT01288911
Title: A Randomized, Double-Blind, Phase II, Efficacy and Safety Study of MDV3100 Versus Bicalutamide in Castrate Men With Metastatic Prostate Cancer
Brief Title: A Study of Enzalutamide Versus Bicalutamide in Castrate Men With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9785-CL-0222; 2010-021868-15 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Neoplasms
Keywords: Metastatic; MDV3100; Prostate; progressive; Cancer; enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — enzalutamide; bicalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enzalutamide (Experimental): Participants received enzalutamide 160 mg orally once daily until confirmed radiographic disease progression, skeletal-related event or the initiation of a new antineoplastic therapy.
  Interventions: Drug: enzalutamide
- Bicalutamide (Active Comparator): Participants received bicalutamide 50 mg orally once daily until confirmed radiographic disease progression, skeletal-related event or the initiation of a new antineoplastic therapy.
  Interventions: Drug: bicalutamide

INTERVENTIONS:
Drug: enzalutamide — capsules
  Other Names: MDV3100
  Arms: Enzalutamide
Drug: bicalutamide — tablets
  Other Names: Casodex
  Arms: Bicalutamide

SUMMARY:
The purpose of this study was to determine the efficacy and safety of oral enzalutamide compared to bicalutamide in castrate men with metastatic prostate cancer who have progressed while on Luteinizing Hormone Receptor Hormone (LHRH) agonist/antagonist or after receiving a bilateral orchiectomy.

DETAILED DESCRIPTION:
An open-label period was added to the main protocol. Following unblinding at the end of the double-blind period and demonstration of a statistically significant advantage of enzalutamide over bicalutamide as assessed by the primary endpoint, all ongoing enzalutamide treated participants and ongoing or previous bicalutamide treated participants that met entry criteria were offered open-label enzalutamide at the discretion of the participant and study investigators.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Ongoing androgen deprivation therapy with a Luteinizing Hormone Receptor Hormone (LHRH) agonist or antagonist at a stable dose and schedule within 4 weeks of randomization or bilateral orchiectomy (i.e., surgical or medical castration)
* Metastatic disease documented by one of the following:

  * At least two bone lesions on bone scan, or
  * Soft tissue disease documented by computed tomography (CT)/ magnetic resonance imaging (MRI), or
  * Unequivocal pelvic adenopathy short axis > 2.0 cm in diameter by CT/MRI
* Progressive disease at study entry defined as one or more of the following three criteria occurring in the setting of castrate levels of testosterone:

  * Prostate Specific Antigen (PSA) progression defined by a minimum of three rising PSA levels with an interval of ≥ 1 week between each determination. The PSA value should be ≥ 2 µg/L (2 ng/mL);
  * Soft tissue disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
  * Bone disease progression defined by two or more new lesions on bone scan
* Asymptomatic or mildly symptomatic from prostate cancer (i.e. the score on the Brief Pain Inventory-Short Form (BPI-SF) Question #3 must be < 4); no use of opiate analgesics for prostate cancer-related pain currently or anytime within 4 weeks prior to randomization
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, including subjects with decreased performance status not attributed to progressive and symptomatic prostate cancer
* Estimated life expectancy of ≥ 12 months
* Able to swallow the study drug and comply with study requirements
* A male subject and his female spouse/partner who is of childbearing potential must use two acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at Screening and continuing throughout the study period, and for 3 months after final study drug administration. Two acceptable forms of birth control include:

  1. Condom (barrier method of contraception), AND
  2. In addition to a condom, one of the following acceptable forms of contraception is required:

     * Established use of oral, injected or implanted hormonal methods of contraception.
     * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
     * Barrier methods of contraception: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
     * Tubal ligation for at least 6 months prior to Screening
     * Vasectomy or other surgical castration at least 6 months prior to Screening

Exclusion Criteria:

* Prior cytotoxic chemotherapy for prostate cancer
* Severe concurrent disease, infection, or comorbidity that would make the subject inappropriate for enrollment
* Known or suspected brain and/or skull metastasis or active epidural disease
* History of another malignancy within the previous 5 years other than curatively treated non-melanomatous skin cancer
* Current or prior treatment with estrogens and/or drugs with anti-androgenic properties such as spironolactone > 50 mg/day, or progestational agents for the treatment of prostate cancer within 6 months prior to randomization
* Current or prior use of ketoconazole for the treatment of prostate cancer
* Use of antiandrogens within 6 weeks prior to randomization
* Documented prior disease progression while receiving antiandrogens. Disease progression defined as PSA progression, radiographic progression and/or clinical deterioration.
* Current or prior treatment with 5-α reductase inhibitors or anabolic steroids within 6 months prior to randomization
* Prior use of systemic glucocorticoids (the equivalent of 10 mg of prednisone) within 3 months prior to randomization or expectation of their use during the study
* Radiation therapy to bone lesions or prostatic bed within 4 weeks prior to randomization
* Major surgery within 2 months prior to randomization
* History of seizure including febrile seizure or any condition that may predispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization). Also, current or prior treatment with anti-epileptic medications for the treatment of seizures or history of loss of consciousness or transient ischemic attack within 12 months prior to randomization
* Clinically significant cardiovascular disease including myocardial infarction within past six months or uncontrolled angina within past three months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2011-03-22 (Actual); Primary Completion 2014-10-19 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Carolina Urologic Research Center; Associate Medical Science Director, Study Director — Astellas Pharma Global Development
Locations (88):
- United States (36):
  - Site US1934, Homewood, Alabama
  - Site US1527, Anchorage, Alaska
  - Site US3026, Tucson, Arizona
  - Site US2977, Highland, California
  - Site US3630, San Diego, California
  - Site US2935, Denver, Colorado
  - Site US2945, Middlebury, Connecticut
  - Site US2014, Melrose Park, Illinois
  - Site US2067, Springfield, Illinois
  - Site US2027, Jeffersonville, Indiana
  - Site US1838, West Des Moines, Iowa
  - Site US62, Kansas City, Kansas
  - Site US2976, Baltimore, Maryland
  - Site US3182, Bethesda, Maryland
  - Site US2975, Ann Arbor, Michigan
  - Site US892, Grand Rapids, Michigan
  - Site US20, Minneapolis, Minnesota
  - Site US3078, Billings, Montana
  - Site US2968, Lawrenceville, New Jersey
  - Site US3025, Poughkeepsie, New York
  - Site US1675, Rochester, New York
  - Site US2934, Staten Island, New York
  - Site US81, Chapel Hill, North Carolina
  - Site US2104, Greensboro, North Carolina
  - Site US44, Cincinnati, Ohio
  - Site US2185, Columbus, Ohio
  - Site US1598, Bala-Cynwyd, Pennsylvania
  - Site US1680, Lancaster, Pennsylvania
  - Site US2926, Myrtle Beach, South Carolina
  - Site US1657, Nashville, Tennessee
  - Site US464, Houston, Texas
  - Site US2978, San Antonio, Texas
  - Site US1653, Virginia Beach, Virginia
  - Site US1580, Burien, Washington
  - Site US1709, Wenatchee, Washington
  - Site US51, Milwaukee, Wisconsin
- Belgium (6):
  - Site BE3015, Brussels
  - Site BE1322, Ghent
  - Site BE3018, Kortrijk
  - Site BE3288, Leuven
  - Site BE3289, Liège
  - Site BE3013, Turnhout
- Canada (7):
  - Site CA3104, Calgary, Alberta
  - Site CA3242, Abbotsford, British Columbia
  - Site CA2646, Kingston, Ontario
  - Site CA166, Toronto, Ontario
  - Site CA3084, Toronto, Ontario
  - Site CA2984, Granby, Quebec
  - Site CA170, Montreal, Quebec
- Denmark (4):
  - Site DK3354, Aalborg
  - Site DK3356, Aarhus
  - Site DK1857, Copenhagen
  - Site DK1263, Herlev
- France (8):
  - Site FR1091, Créteil
  - Site FR3009, Lille
  - Site FR442, Lyon
  - Site FR3002, Paris
  - Site FR3003, Poitiers
  - Site FR3000, Rennes
  - Site FR3007, Rouen
  - Site FR3005, Suresnes
- Germany (11):
  - Site DE4000, Nürtingen, Baden-Wurttemberg
  - Site DE2989, Aachen
  - Site DE3287, Bergisch Gladbach
  - Site DE2993, Bonn
  - Site DE2995, Bonn
  - Site DE2994, Bonn
  - Site DE2990, Hamburg
  - Site DE3270, Hanover
  - Site DE2992, Reutlingen
  - Site DE3286, Waldshut-Tiengen
  - Site DE2988, Wuppertal
- Romania (3):
  - Site RO3042, Bucharest, RO
  - Site RO3039, Bucharest, RO
  - Site RO3035, Bucharest
- United Kingdom (13):
  - Site GB3029, Bristol, UK
  - Site GB3027, London, UK
  - Site GB3030, London, UK
  - Site GB3028, Cardiff, Wales
  - Site GB3244, Belfast
  - Site GB2702, Cambridge
  - Site GB3166, Glasgow
  - Site GB1862, Leicher
  - Site GB3163, London
  - Site GB2624, Manchester
  - Site GB3355, Merseyside
  - Site GB3245, Northwood, Middlesex
  - Site GB3290, Preston

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Schultz NM, Shore ND, Chowdhury S, Klotz LH, Concepcion RS, Penson DF, Karsh LI, Yang H, Brown BA, Barlev A, Flanders SC. Number-needed-to-treat analysis of clinical progression in patients with metastatic castration-resistant prostate cancer in the STRIVE and TERRAIN trials. BMC Urol. 2018 Sep 6;18(1):77. doi: 10.1186/s12894-018-0387-7. PMID 30189902
- [Derived] Heidenreich A, Chowdhury S, Klotz L, Siemens DR, Villers A, Ivanescu C, Holmstrom S, Baron B, Wang F, Lin P, Shore ND. Impact of Enzalutamide Compared with Bicalutamide on Quality of Life in Men with Metastatic Castration-resistant Prostate Cancer: Additional Analyses from the TERRAIN Randomised Clinical Trial. Eur Urol. 2017 Apr;71(4):534-542. doi: 10.1016/j.eururo.2016.07.027. Epub 2016 Aug 3. PMID 27497762
- [Derived] Shore ND, Chowdhury S, Villers A, Klotz L, Siemens DR, Phung D, van Os S, Hasabou N, Wang F, Bhattacharya S, Heidenreich A. Efficacy and safety of enzalutamide versus bicalutamide for patients with metastatic prostate cancer (TERRAIN): a randomised, double-blind, phase 2 study. Lancet Oncol. 2016 Feb;17(2):153-163. doi: 10.1016/S1470-2045(15)00518-5. Epub 2016 Jan 14. PMID 26774508
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=282

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men with metastatic castration-resistant prostate cancer (mCRPC) were enrolled at 84 sites in a total of 8 countries.
Pre-assignment Details: Participants were stratified by whether bilateral orchiectomy or receipt of luteinizing hormone-releasing hormone (LHRH) agonist/antagonist therapy started before or after the diagnosis of metastases and by site.
Period: Double-blind Period
Arm/Group | Enzalutamide | Bicalutamide
Started | 184 | 191
Received Treatment | 183 | 189
Completed | 42 (Indicates participants were still receiving treatment at the data cut-off date of 19 October 2014.) | 9 (Indicates participants were still receiving treatment at the data cut-off date of 19 October 2014.)
Not Completed | 142 | 182
Not completed — Death | 11 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Progressive Disease | 75 | 103
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 25 | 26
Not completed — Miscellaneous Reason | 29 | 42
Not completed — Randomized but never received study drug | 1 | 2
Period: Open-label Period (All Enzalutamide)
Arm/Group | Enzalutamide | Bicalutamide
Started | 42 | 9
Received Treatment | 42 | 9
Completed | 0 | 0
Not Completed | 42 | 9
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Progressive disease | 18 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Miscellaneous Reason | 5 | 0
Not completed — Transitioned to 9785-CL-0123 NCT02960022 | 17 | 5

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all participants that were randomized to receive study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzalutamide | Bicalutamide | Total
Number analyzed (Participants) | 184 | 191 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (9.22) | 71.1 (8.89) | 70.7 (9.05)
Age, Customized [Number; unit: participants]
  < 65 years | 45 | 47 | 92
  65-75 years | 85 | 80 | 165
  > 75 years | 54 | 64 | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 184 | 191 | 375
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 172 | 176 | 348
  Black or African American | 8 | 10 | 18
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Other | 0 | 2 | 2
Ethnicity [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 184 | 187 | 371
  Hispanic or Latino | 0 | 4 | 4
LHRH agonist/antagonist initiation or bilateral orchiectomy relative to diagnosis of metastasis [Count of Participants; unit: Participants]
  Before diagnosis of metastasis | 87 | 76 | 163
  After diagnosis of metastasis | 97 | 115 | 212

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Independent Central Review (ICR) Assessment
Description: PFS is the time from randomization to the date of the first progression event detected. A progression event was defined as objective evidence of radiographic disease progression based on the assessments by the ICR, skeletal-related event, initiation of new antineoplastic therapy or death by any cause, whichever occurred first. Radiographic disease progression was defined as either a progression in soft tissue on computed tomography (CT)/magnetic resonance imaging (MRI) scan according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, and/or a progression in bone lesions on bone scan (≥ 2 new bone lesions) confirmed by the next bone scan. A skeletal-related event was any radiation therapy or surgery to bone, pathologic bone fracture, spinal cord compression or change in antineoplastic therapy to treat bone pain. The initiation of new antineoplastic therapy included any new therapy for the treatment of disease progression after the study drug administration started.
Time Frame: From randomization until the data cut-off date of 19 October 2014, median duration of treatment was 11.6 months in the enzalutamide arm and 5.8 months in the bicalutamide arm.
Population: Full analysis set (all randomized participants)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
months | 15.7 [11.5 to 19.4] | 5.8 [4.8 to 8.1]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; PFS based on ICR Enzalutamide Vs. Bicalutamide. The (unstratified) log-rank test with an overall significance level of 0.05 (two-sided) was used to compare the PFS of enzalutamide to bicalutamide. The (unstratified) Cox proportional hazards model was used to estimate the hazard ratio of enzalutamide to bicalutamide, calculate the corresponding two-sided 95% confidence intervals and test the hypothesis that the hazard ratio is equal to 1; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.34 to 0.57] — Estimated by use of Cox proportional hazards model

2. Secondary Outcome: PFS Based on Investigator Assessment
Description: PFS was calculated as the time from randomization to the date of the first progression event detected. A progression event was defined as objective evidence of radiographic disease progression based on the assessments by investigators, skeletal-related event, initiation of new antineoplastic therapy or death by any cause, whichever occurred first. Radiographic disease progression was defined as either a progression in soft tissue on CT/MRI scan according to RECIST 1.1, and/or a progression in bone lesions on bone scan (≥ 2 new bone lesions) confirmed by the next bone scan. A skeletal-related event was defined as radiation therapy or surgery to bone, pathologic bone fracture, spinal cord compression or change in antineoplastic therapy to treat bone pain. The initiation of new antineoplastic therapy included any new therapy for the treatment of disease progression after the study drug administration started.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
months | 15.3 [11.8 to 19.4] | 5.7 [5.4 to 8.1]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; PFS on based investigator assessment Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.33 to 0.55] — Estimated by use of Cox proportional hazards model

3. Secondary Outcome: Prostate-specific Antigen (PSA) Response by Week 13
Description: The PSA response by Week 13 was defined as the percentage change from Baseline to the smallest PSA value after Baseline (i.e., a decrease of 100% represents the largest possible decrease to a value below the lower limit of quantification) and on or before day 99 (i.e., upper boundary of the Week 13 visit window). For participants with no decrease in PSA post-baseline by Week 13, the PSA response by Week 13 was the smallest increase in PSA up to day 99. For participants with no post-baseline PSA values up to day 99, the PSA response by Week 13 was set to missing. PSA was analyzed at a central laboratory.
Time Frame: Baseline to Week 13
Population: Full analysis set with available PSA data
Measure: Median (Full Range); unit: percent change
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 171 | 163
percent change | -89.03 [-100.0 to 287.7] | 0.36 [-98.5 to 25700.0]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; PSA Response Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test

4. Secondary Outcome: Best PSA Response
Description: The best PSA response was defined as the percentage change from Baseline to the smallest PSA value after Baseline including PSA results from samples taken after the study drug was stopped. For participants with no decrease in PSA post-baseline, the best PSA response was the smallest increase in PSA. For participants with no post-baseline PSA values, the PSA response was set to missing. PSA was analyzed at a central laboratory.
Time Frame: Baseline to the data cutoff date of 19 October 2014, median duration of treatment was 11.6 months in the enzalutamide arm and 5.8 months in the bicalutamide arm.
Population: Full analysis set with available PSA data
Measure: Median (Full Range); unit: percent change
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 174 | 168
percent change | -92.96 [-100.0 to 287.7] | 0.18 [-99.8 to 25700.0]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Best PSA Response Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test

5. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was calculated as the time interval from the date of randomization to the date of first observation of PSA progression. PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir (or above the baseline value for participants who did not have a decline in PSA post-baseline values), and confirmed by a second consecutive PSA assessment at least 3 weeks later. For participants with no documented PSA progression, the time to PSA progression was censored on the date the last PSA sample was taken.
Time Frame: From randomization until the data cutoff date of 19 October 2014, median duration of treatment was 11.6 months in the enzalutamide arm and 5.8 months in the bicalutamide arm.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
months | 19.4 [16.6 to NA] — Not reached due to the low number of events | 5.8 [5.6 to 8.3]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Time to PSA progression Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.20 to 0.39] — Estimated by use of Cox proportional hazards model

6. Secondary Outcome: Time to PSA ≤ 4 ng/mL
Description: Time to PSA ≤ 4 ng/mL was defined as the time interval from the date of randomization to the first date a decline in PSA to a result of 4 ng/mL or below was recorded. In participants without PSA results ≤ 4 ng/mL, the time to PSA ≤ 4 ng/mL was censored on the date of the last PSA sample taken. Participants with a PSA result ≤ 4 ng/mL at Baseline, participants with no Baseline PSA and participants with no post-baseline PSA results were censored on the date of randomization
Time Frame: as for outcome 5
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
months | 3.0 [2.9 to 5.6] | NA [NA to NA] — Not reached due to the low number of events
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Time to PSA Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 5.07, 95% CI 2-sided [3.18 to 8.09] — Estimated by use of Cox proportional hazards model

7. Secondary Outcome: Time to ≥ 30% PSA Decline From Baseline
Description: The time to ≥ 30% PSA decline from Baseline was defined as the time interval from the date of randomization to the first date a PSA decline from Baseline of at least 30% was recorded. In participants without ≥ 30% PSA decline from Baseline, the time to ≥ 30% PSA decline from Baseline was censored on the date of the last PSA sample taken. Participants who had no Baseline PSA and participants with no post-baseline PSA results were censored on the date of randomization.
Time Frame: as for outcome 5
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
months | 2.8 [2.8 to 2.8] | NA [NA to NA] — Not reached due to the low number of events
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Time to ≥ 30% PSA decline from baseline Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 5.55, 95% CI 2-sided [3.96 to 7.79] — Estimated by use of Cox proportional hazards model

8. Secondary Outcome: Time to ≥ 50% PSA Decline From Baseline
Description: The time to ≥ 50% PSA decline from Baseline was defined as the time interval from the date of randomization to the first date a PSA decline from Baseline of at least 50% was recorded. In participants without ≥ 50% PSA decline from Baseline, the time to ≥ 50% PSA decline from Baseline was censored on the date of the last PSA sample taken. Participants who had no Baseline PSA and participants with no post-baseline PSA results were censored on the date of randomization.
Time Frame: as for outcome 5
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
months | 2.8 [2.8 to 2.8] | NA [NA to NA] — Not reached due to the low number of events
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Time to ≥ 50% PSA decline from baseline Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 7.01, 95% CI 2-sided [4.83 to 10.16] — Estimated by use of Cox proportional hazards model

9. Secondary Outcome: Time to ≥ 90% PSA Decline From Baseline
Description: The time to ≥ 90% PSA decline from Baseline was defined as the time interval from the date of randomization to the first date a PSA decline from Baseline of at least 90% was recorded. In participants without ≥ 90% PSA decline from Baseline, the time to ≥ 90% PSA decline from Baseline was censored on the date of the last PSA sample taken. Participants who had no Baseline PSA and participants with no post-baseline PSA results were censored on the date of randomization.
Time Frame: as for outcome 5
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
months | 5.4 [3.0 to 5.7] | NA [NA to NA] — Not reached due to the low number of events
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Time to ≥ 90% PSA decline from baseline Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 13.91, 95% CI 2-sided [7.23 to 26.79] — Estimated by use of Cox proportional hazards model

10. Secondary Outcome: Radiographic PFS Based on ICR Assessment
Description: Radiographic PFS was calculated as the time interval from the date of randomization to the first date of radiographic disease progression. Radiographic disease progression was defined as either a progression in soft tissue on CT/MRI scan according to RECIST 1.1, and/or a progression in bone lesions (a minimum of 2 new bone lesions as compared to previous scan) on bone scan and confirmed by the next bone scan.
Time Frame: as for outcome 5
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
months | NA [25.6 to NA] — Not reached due to the low number of events | 16.4 [11.1 to 18.1]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Radiographic PFS based on ICR Enzalutamide Vs. Bicalutamide; Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.36 to 0.74] — Estimated by use of Cox proportional hazards model

11. Secondary Outcome: Percentage of Participants With an Objective Response
Description: Response assessments were reported by ICR for target lesions in soft tissues and non-target lesions in soft tissues based on CT and/or MRI according to RECIST version 1.1. Objective response was defined as the number of participants achieving either a complete response (CR) or a partial response (PR) based on participant's best overall response assessed at the end of the treatment.
Time Frame: as for outcome 5
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 184 | 191
percentage of participants | 15.8 | 2.6

12. Secondary Outcome: Percentage of Participants With Adverse Events
Description: A serious adverse event was defined as any untoward medical occurrence that at any dose: ● Resulted in death ● Was life threatening ● Resulted in persistent or significant disability/incapacity ● Resulted in congenital anomaly or birth defect ● Required inpatient hospitalization or led to prolongation of hospitalization ● Other medically important events. Treatment-related indicates adverse events assessed by the Investigator as probably or possibly related to study treatment. Treatment emergent adverse events (TEAEs) were defined as adverse events (AEs) that started or worsened after starting administration of study drug through end of the study (i.e., the treatment-emergent period).
Time Frame: From initiation of study drug up to 30 days after last dose of study drug or the 30-day safety follow-up visit, whichever was last (Median duration of treatment was 11.6 months in enzalutamide arm and 5.8 in bicalutamide arm, 12.6 in the total arm).
Population: Safety Analysis Set (all participants who had initiated at least 1 dose of study drug)
Measure: Number; unit: percentage of participants
Groups:
- Total Enzalutamide: Participants received enzalutamide in the double-blind and/or open-label period (including participants who switched from bicalutamide to enzalutamide).
Arm/Group | Enzalutamide | Bicalutamide | Total Enzalutamide
Number analyzed (Participants) | 183 | 189 | 192
percentage of participants
  TEAEs | 94.5 | 94.2 | 94.8
  Related TEAEs | 66.7 | 49.7 | 67.2
  Deaths | 5.5 | 1.6 | 5.7
  Serious TEAEs | 33.3 | 23.8 | 36.5
  Drug regimen-related serious TEAEs | 6.6 | 3.2 | 6.8
  TEAEs leading to discontinuation | 29.5 | 23.8 | 31.3
  Drug regimen-related TEAEs leading to discon. | 7.7 | 5.3 | 7.8
  TEAEs leading to study drug interruption | 10.4 | 7.9 | 10.4

ADVERSE EVENTS:
Time Frame: From initiation of study drug up to 30 days after the last dose of study drug or the 30-day safety follow-up visit, whichever occurred last. Median duration of treatment was 11.6 months in the enzalutamide arm and 5.8 months in the bicalutamide arm in the double-blind period. In the open-label period, the median duration of treatment was 21.6 months in participants who previously received enzalutamide and 20.9 months in participants who previously received bicalutamide.
Description: The total number of deaths (all causes) includes deaths reported after the time frame above.
Groups:
- Double-blind Period: Enzalutamide: Participants received enzalutamide 160 mg orally once daily in the double-blind period until confirmed radiographic disease progression, skeletal-related event or the initiation of a new antineoplastic therapy.
- Double-blind Period: Bicalutamide: Participants received bicalutamide 50 mg orally once daily in the double-blind period until confirmed radiographic disease progression, skeletal-related event or the initiation of a new antineoplastic therapy.
- Open-label Period: Enzalutamide/Enzalutamide: Participants received enzalutamide in the double-blind period and received enzalutamide in the open-label period as well.
- Open-label Period: Bicalutamide/Enzalutamide: Participants received bicalutamide in the double-blind period and switched over to enzalutamide in the open-label period.
Arm/Group | Double-blind Period: Enzalutamide | Double-blind Period: Bicalutamide | Open-label Period: Enzalutamide/Enzalutamide | Open-label Period: Bicalutamide/Enzalutamide
All-Cause Mortality (participants affected / at risk) | 11/141 | 7/180 | 0/42 | 1/9
Serious Adverse Events (participants affected / at risk) | 49/141 | 43/180 | 18/42 | 4/9
Other Adverse Events (participants affected / at risk) | 123/141 | 149/180 | 42/42 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Period: Enzalutamide (N=141) | Double-blind Period: Bicalutamide (N=180) | Open-label Period: Enzalutamide/Enzalutamide (N=42) | Open-label Period: Bicalutamide/Enzalutamide (N=9)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess of salivary gland (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epiduritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incoherent (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (4) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Period: Enzalutamide (N=141) | Double-blind Period: Bicalutamide (N=180) | Open-label Period: Enzalutamide/Enzalutamide (N=42) | Open-label Period: Bicalutamide/Enzalutamide (N=9)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 5 (7) | 4 (4) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 7 (7) | 3 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 19 (21) | 24 (25) | 5 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 16 (18) | 15 (18) | 5 (6) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 4 (4) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (22) | 33 (36) | 10 (11) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 9 (10) | 1 (1) | 0 (0)
Asthenia (General disorders) | 8 (10) | 7 (7) | 2 (2) | 0 (0)
Fatigue (General disorders) | 35 (40) | 38 (45) | 18 (24) | 3 (3)
Oedema peripheral (General disorders) | 10 (10) | 13 (13) | 5 (5) | 0 (0)
Pain (General disorders) | 1 (1) | 8 (8) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 4 (4) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (13) | 7 (8) | 7 (9) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 7 (8) | 3 (3) | 4 (4) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 9 (11) | 6 (7) | 4 (6) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 3 (4) | 5 (6) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (4) | 5 (5) | 1 (1) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Red blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 16 (19) | 15 (15) | 5 (6) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 16 (19) | 13 (13) | 2 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (22) | 27 (39) | 9 (11) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (39) | 34 (40) | 11 (15) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 12 (15) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 3 (3) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 4 (4) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 17 (23) | 5 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (5) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 4 (4) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (22) | 9 (12) | 5 (8) | 1 (1)
Amnesia (Nervous system disorders) | 4 (5) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 12 (15) | 15 (16) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 11 (14) | 6 (6) | 8 (10) | 3 (4)
Lethargy (Nervous system disorders) | 5 (6) | 4 (4) | 3 (3) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 9 (9) | 8 (8) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 5 (5) | 4 (4) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (5) | 6 (7) | 5 (5) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 7 (7) | 6 (6) | 1 (1) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 5 (7) | 1 (1) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 4 (4) | 2 (2) | 6 (6) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (8) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 9 (10) | 4 (8) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Jaw operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 15 (16) | 17 (17) | 12 (12) | 4 (5)
Hypertension (Vascular disorders) | 18 (29) | 14 (16) | 13 (16) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.